CLINICAL TRIAL: NCT05806112
Title: Effectiveness of Interventions to Improve Resiliency & Burnout in Behavioral Health Residential Staff
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Vinfen (Industry); Bay Cove Human Services (Other)
Responsible Party: Principal Investigator, Stephen Bartels, Director of the Mongan Institute at Massachusetts General Hospital, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2023P000476
Record Dates: First submitted 2023-03-27; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Burnout; Stress; Coping Skills; Depression; Anxiety; Physical Inactivity; Sleep; Healthy Eating
Keywords: group home; resiliency; residential care worker; burnout; turnover
MeSH Terms: conditions — Burnout, Psychological; Depression; Anxiety Disorders; Sedentary Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated Resiliency Training and Task Sharing (Experimental): A multi-component intervention combining resiliency training and task sharing implemented at the site-level (microsystem).
  Interventions: Behavioral: Resiliency Training; Behavioral: Task Sharing
- Workplace Improvement Learning Collaborative (Experimental): A workplace improvement learning collaborative implemented at the organization level (mesosystem).
  Interventions: Behavioral: Workplace Improvement Learning Collaborative

INTERVENTIONS:
Behavioral: Resiliency Training — The Stress Management and Resiliency Training: Relaxation Response Resiliency Program (SMART-3RP) has been shown to be effective in improving resilience and reducing distress among individuals across different populations and settings. The SMART-3RP enhances resilience by 1) teaching tools to elicit the relaxation response (RR) to offset negative effects of chronic stress; 2) improving stress management and awareness; and 3) promoting growth enhancement and agency to effect positive change. It blends stress coping principles from mind-body, cognitive-behavioral, and positive psychology theory to teach skills to advance each of these resiliency processes. The training will be delivered in six 50-minute virtual group sessions with 2 optional "booster sessions" available for those who desire additional sessions to further consolidate the core resiliency skills.
  Other Names: The Stress Management and Resiliency Training: Relaxation Response Resiliency Program; SMART-3RP
  Arms: Integrated Resiliency Training and Task Sharing
Behavioral: Task Sharing — Task Sharing is a process involving health care workers in partnership with others in which workers retain many of their primary tasks, but some tasks are completed collaboratively or by other workers or volunteers in a shared effort. Study coaches will work with the group home directors and RCWs to identify shared tasks that may be conducted by peers or resident volunteers by task co-assignment with supervision and support. Task co-assignments will be discussed in routine house meetings occurring on a weekly basis and incorporated into a jointly developed "house plan". The house plan will engage staff and residents to identify shared activities to reduce the burden on RCWs through task co-assignment and team-based efforts aimed at tasks that create unnecessary burden and stress for RCWs, yet do not require RCWs to complete them.
  Arms: Integrated Resiliency Training and Task Sharing
Behavioral: Workplace Improvement Learning Collaborative — The Workplace Improvement Learning Collaborative (WILC) consists of identifying major sources of RCW burnout across the system and then instituting an organizational (agency-wide) measure to address the identified sources of burnout by restructuring tasks (e.g., reducing administrative burdens, increasing workflow efficiencies) through a virtual earning collaborative with group home leaders. Learning collaboratives commonly use a structured framework within which teams learn about research and best practices, apply quality-improvement methods, and exchange their experiences in making improvements with the widespread use of such collaboratives. Program Directors will participate in a learning collaborative facilitated by trained and certified study coaches to identify and collaboratively develop and implement effective strategies to address root causes of RCW burnout across group homes and program directors assigned to the WILC intervention.
  Arms: Workplace Improvement Learning Collaborative

SUMMARY:
The goal of this clinical trial is to compare Integrated Resiliency Training and Task Sharing (IRTTS) to Workplace Improvement Learning Collaborative (WILC) in group homes for adults with serious mental illness and/or intellectual and developmental disabilities. The main questions it aims to answer are:

* Is IRTTS superior to WILC in improving residential care worker (RCW) resiliency; stress management and burnout; depression and anxiety; and positive health behaviors?
* Is IRTTS superior to WILC in improving RCW turnover/retention; RCW sick days/absenteeism; and group home safety and resident incidents?
* What are the barriers, facilitators, and resources required to successfully implement IRTTS and WILC?

Participants may engage in training sessions, collaborate with residents and other RCWs in their group homes, attend meetings with RCWs from other group homes, complete surveys, participate in focus groups, and/or give qualitative interviews.

Researchers will compare IRTTS to WILC to see which intervention should be implemented to achieve the greatest improvement in RCW resiliency and greatest reduction in burnout and turnover in group homes for adults with serious mental illness and/or developmental and intellectual disabilities.

DETAILED DESCRIPTION:
This study involves group homes for adults (age 18+) with serious mental illness (DSM-V Diagnosis of Axis-I Mental Illness with persistent functional impairment) and group homes for adults with developmental and intellectual disabilities operated by public-sector community-based human service organizations. Approximately n=180 group homes operated by two human services organizations in Massachusetts (Vinfen and Bay Cove Human Services) with approximately 900 residential care workers (RCWs) will be included in this study.

To test whether site-level Integrated Resiliency Training and Task Sharing (IRTTS) is superior to an organization-level Workplace Improvement Learning Collaborative (WILC) in improving RCW-level and group-home-level outcomes, researchers will conduct a cluster randomized trial randomizing n=180 congregate care homes to either IRTTS (n=90 homes) or WILC (n=90 homes) in three 18-month phases over the study period (60 homes enrolled per phase). Note: the unit of randomization is group home, not individual RCW. Cluster randomization is adopted as the interventions are system-level interventions delivered to groups of individuals in each home. As IRTTS consists of training RCWs in group-based resiliency, researchers will provide training to approximately 5 RCWs in each group home and evaluate outcomes for 90 group homes and approximately 450 RCWs assigned to IRTTS (30 IRTTS group homes and 150 IRTTS RCWs in each of three phases of the implementation). WILC consists of a learning collaborative approach involving group home leaders. For the n=90 WILC group homes, researchers will involve n=90 group home leaders and will evaluate the impact on group home-level outcomes for the n=90 group homes on approximately 450 RCWs assigned to WILC (30 WILC group homes and 150 WILC RCWs in each of the three phases of implementation). The project will take place over four years.

ELIGIBILITY:
Inclusion Criteria:

* Permanent-salary staff working in participating group homes

Exclusion Criteria:

* Temp staff and per diem workers
* Staff working in group homes not included in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Resilience (baseline) | Baseline
  Resilience is assessed using the Current Experiences Scale (CES). The CES is a 23-item measure with total scores that can range from 0 to 115, with higher scores indicating greater resiliency.
Resilience (3-month follow-up) | 3-months
  Resilience is assessed using the Current Experiences Scale (CES). The CES is a 23-item measure with total scores that can range from 0 to 115, with higher scores indicating greater resiliency.
Resilience (12-month follow-up) | 12-months
  Resilience is assessed using the Current Experiences Scale (CES). The CES is a 23-item measure with total scores that can range from 0 to 115, with higher scores indicating greater resiliency.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No